CLINICAL TRIAL: NCT02535117
Title: Laparoscopic Surgery Versus Radiofrequency Ablation for Recurrent Hepatocellular Carcinoma After Initial Partial Hepatectomy: A Multicenter Experience
Brief Title: Laparoscopic Surgery Versus Radiofrequency Ablation for Recurrent HCC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhen-Wei Peng, Ph.D.,M.D., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 003
Record Dates: First submitted 2015-08-24; First posted 2015-08-28 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Surgery(LS) (Experimental): For LS, the patient was usually placed in the lithotomy position. Pneumoperitoneum was maintained at a pressure between 12 and 14 mmHg. Three to 4 working ports sized between 5 mm and 12 mm were used . Intra-operative ultrasonography was performed routinely. Parenchymal transection was performed using a Cavitron ultrasonic surgical aspirator (CUSA, Valleylab, Boulder, CO, USA). Large bile duct branches or vessels were clipped before division and minor hemostasis was carried out using bipolar diathermy. Large hepatic vein branches were divided by endovascular staplers. A 1.0-cm safety margin was planed to get during the liver resection.
  Interventions: Procedure: Laparoscopic Surgery(LS)
- RFA (Active Comparator): RFA was performed according to the Guidelines of Radiofrequency Ablation Therapy for Liver Cancer: Chinese Expert Consensus Statement issued by the Chinese Society of Liver Cancer and Chinese Society of Clinical Oncology RFA was performed under real-time ultrasound guidance. RFA was performed by using a commercially available Cool-tipTM RFA system (Valleylab, Boulder, CO, USA), or a RF 2000 system (Radio-Therapeutics Mountain View, CA). Grounding was achieved by attaching 2 pads to the patient's back or legs.
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: Laparoscopic Surgery(LS) — For LS, the patient was usually placed in the lithotomy position. Pneumoperitoneum was maintained at a pressure between 12 and 14 mmHg. Three to 4 working ports sized between 5 mm and 12 mm were used . Intra-operative ultrasonography was performed routinely. Parenchymal transection was performed using a Cavitron ultrasonic surgical aspirator (CUSA, Valleylab, Boulder, CO, USA). Large bile duct branches or vessels were clipped before division and minor hemostasis was carried out using bipolar diathermy. Large hepatic vein branches were divided by endovascular staplers. A 1.0-cm safety margin was planed to get during the liver resection.
  Arms: Laparoscopic Surgery(LS)
Procedure: RFA — RFA was performed according to the Guidelines of Radiofrequency Ablation Therapy for Liver Cancer: Chinese Expert Consensus Statement issued by the Chinese Society of Liver Cancer and Chinese Society of Clinical Oncology RFA was performed under real-time ultrasound guidance. RFA was performed by using a commercially available Cool-tipTM RFA system (Valleylab, Boulder, CO, USA), or a RF 2000 system (Radio-Therapeutics Mountain View, CA). Grounding was achieved by attaching 2 pads to the patient's back or legs.
  Arms: RFA

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common and the third leading cause of death from cancer worldwide1 . Hepatectomy is still the main effective treatment for HCC accompanying with well-preserved cirrhosis when liver transplantation is not feasible due to the lack of donors Recurrence of tumor within the liver remnant is also common, with a reported 5-year recurrence rate of 50-70%, in patients who have undergone "curative" hepatectomy. Management of recurrent HCC is still urgent and several treatments have been developed. Repeat hepatectomy is considered to be the first choice for recurrent HCC with a 5-year survival rate of 19.4 to 56%. Unfortunately, repeat hepatectomy can be performed only in a small proportion of patients with HCC recurrence due to the poor functional liver reserve or because of widespread recurrence. With a 3-year survival rate of 62% to 68% after treatment, radiofreqency ablation (RFA) has been used as an effective treatment for recurrent HCC. The efficacy of RFA for recurrent HCC has been reported to be comparable to those achieved by surgery. Laparoscopic surgery was considered not to be a suitable treatment for recurrent HCC due to postoperative adhesions that can make laparoscopic surgical procedure more difficult and less safe. Recently, several studies reported that laparoscopic surgery for recurrent HCC in cirrhotic patients is a safe and feasible procedure with good short-term outcomes. By far, no study has been performed to compare the efficacy and safety of laparoscopic surgery with RFA for treatment of recurrent HCC.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years;
2. recurrent HCC after curative partial hepatectomy;
3. no other treatment received except for partial hepatectomy;
4. a solitary recurrent HCC ≤ 5.0 cm in diameter, or multiple recurrent HCC ≤ 3 lesions, each ≤ 3.0 cm in diameter;
5. no radiologic evidence of invasion into major portal/ hepatic vein branches ;
6. no extrahepatic metastases;
7. Child-pugh class A or B liver cirrhosis;
8. American Society of Anesthesiologists (ASA) score ≤ 3;
9. Eastern Co-operative Oncology Group performance (ECOG) status 0;

Exclusion Criteria:

1. coagulation disorders (prothrombin activity <40% or a platelet count of <80,000/mm3);
2. Child-Pugh class C liver cirrhosis;
3. history of hepatic encephalopathy, ascites refractory to diuretics or esophageal or gastric variceal bleeding;
4. a history of a secondary malignancy;
5. active infection (except viral hepatitis);
6. severe dysfunction of the heart, kidney, or other organs

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years

SECONDARY OUTCOMES:
Recurrence-free survival | 5 years
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, Ph.D., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University

REFERENCES:
- [Background] Belli G, Fantini C, D'Agostino A, Cioffi L, Langella S, Russolillo N, Belli A. Laparoscopic versus open liver resection for hepatocellular carcinoma in patients with histologically proven cirrhosis: short- and middle-term results. Surg Endosc. 2007 Nov;21(11):2004-11. doi: 10.1007/s00464-007-9503-6. Epub 2007 Aug 19. PMID 17705086
- [Background] Peng ZW, Zhang YJ, Liang HH, Lin XJ, Guo RP, Chen MS. Recurrent hepatocellular carcinoma treated with sequential transcatheter arterial chemoembolization and RF ablation versus RF ablation alone: a prospective randomized trial. Radiology. 2012 Feb;262(2):689-700. doi: 10.1148/radiol.11110637. Epub 2011 Dec 12. PMID 22157201